CLINICAL TRIAL: NCT05740358
Title: Liver Cirrhosis Network Cohort Study
Acronym: LCN-C
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: The Cleveland Clinic (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); Duke University (Other); Mayo Clinic (Other); University of Miami (Other); University of Michigan (Other); University of California, San Diego (Other); University of California, San Francisco (Other); LAC+USC Medical Center (Other); Virginia Commonwealth University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Cancer Institute (NCI) (NIH); University of Southern California (Other); Central Virginia Veterans Healthcare System (Unknown)
Responsible Party: Principal Investigator, Abigail Smith, Associate Professor, Northwestern University
Other Study IDs: LCN Cohort Study; 1U24DK130164-01 (NIH); Pro00064389 (Other: Advarra, Inc.); 5U01DK130177-02 (NIH); 5U01DK130197-02 (NIH); 5U01DK130185-02 (NIH); 5U01DK130180-02 (NIH); 5U01DK130221-02 (NIH); 5U01DK130134-02 (NIH); 5U01DK130168-02 (NIH); 5U01DK130190-02 (NIH); 5U01DK130113-02 (NIH); 5U01DK130181-02 (NIH); 5U24DK130164-02 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis; Cirrhosis, Liver; Cirrhosis Early; Cirrhosis Due to Hepatitis B; Cirrhosis Advanced; Cirrhosis Infectious; Cirrhosis Alcoholic; Cirrhosis, Biliary; Cirrhosis Cryptogenic; Cirrhosis Due to Hepatitis C; Cirrhosis Due to Primary Sclerosing Cholangitis; Autoimmune Hepatitis
Keywords: Cirrhosis; Liver; Nonalcoholic Fatty Liver Disease; NASH; Nonalcoholic steatohepatitis
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Liver Cirrhosis, Alcoholic; Liver Cirrhosis, Biliary; Cirrhosis, Cryptogenic; Hepatitis, Autoimmune; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, stool (optional)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver Cirrhosis Network (LCN) Cohort Study is an observational study designed to identify risk factors and develop prediction models for risk of decompensation in adults with liver cirrhosis. LCN Cohort Study involves multiple institutions and an anticipated 1200 participants. Enrolled participants will have study visits every 6 months (180 days), with opportunities to complete specific visit components via telehealth or remotely. Visits will include collection of questionnaire data and the in-person visits will include questionnaires, physical exams, imaging, and sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing to provide samples at baseline
* Cirrhosis

Where Cirrhosis is defined as:

1. At least one liver biopsy within 5 years prior to consent showing either: a) Metavir stage 4 fibrosis; Ishak Stage 5-6 fibrosis OR
2. At least 2 of the following:

1. Evidence on imaging: Nodular liver with either splenomegaly or recanalized umbilical vein within the past year 2. Liver stiffness: VCTE within one year prior to consent or during Screening ≥12.5 kPa or MRE within one year prior to consent or during Screening ≥5 kPa 3. Evidence of varices demonstrated on imaging or endoscopy within 3 years prior to consent or during Screening 4. Either: FIB-4>2.67 or platelets <150/mL within 6 months prior to consent or during Screening 5. >5 years METAVIR stage 4 fibrosis or Ishak stage 5-6

Exclusion Criteria:

* Known and documented prior or current hepatocellular carcinoma (HCC) or cholangiocarcinoma
* Known transjugular intrahepatic portosystemic shunt (TIPS), balloon retrograde transvenous obliteration (BRTO) or porto-systemic shunt surgery regardless of time of occurrence
* Known prior solid organ transplant or bone marrow transplant
* Current participation in active medication treatment trials at the time of consent for LCN Cohort Study
* Prisoners or individuals with more than 180 days incarceration pending due to difficulty with visits
* Bariatric surgery in the last 180 days prior to consent
* Known history of fontan procedure-associated liver disease (FALD)
* Known current medical or psychiatric conditions which, in the opinion of the investigator, would make the participant unsuitable for the study or interfere with or prevent follow-up per protocol
* Current liver-unrelated end-stage organ failures (Dialysis, stage 3-4 congestive heart failure (CHF), current chronic obstructive pulmonary disease (COPD) on home oxygen, current known active malignancy besides non-melanomatous skin cancer or carcinoma in situ)
* Documented history of acute alcohol-associated hepatitis (according to NIAAA criteria as described in the MOP) in the 180 days prior to consent
* Documented current or continued signs and symptoms of acute Wilson disease (acute liver failure, acute neurological deficits, hemolysis)
* In patients with primary sclerosing cholangitis (PSC): Current active cholangitis with 90 days prior to consent
* Documented cardiac cirrhosis
* Known recent (within the last 365 days) or present hepatic decompensation with ascites/hydrothorax (including trace ascites discovered at screening not requiring intervention), hepatic encephalopathy or variceal bleeding. If a patient has had a history of decompensation, they must have been off any medications to treat decompensation for at least 365 days. Refer to the MOP for clarifying details on evaluating eligibility for patients with a history of prior decompensation.
* Known or documented habitual non-adherence to previous research studies or medical procedures or unwillingness to adhere to protocol (e.g., unwilling to obtain consent or samples)
* Current model for end-stage liver disease (MELD-Na) cut off ≥ 15*
* Current Child-Turcotte-Pugh (CTP) B or C*
* Current known Hepatitis C Virus (HCV) without sustained virologic response (SVR)
* Current known quantifiable Hepatitis B Virus (HBV) viral DNA on therapy with ongoing adherence on suppressive therapy*
* In patients with autoimmune hepatitis: serum aspartate aminotransferase (AST) > 2X upper limit of normal (ULN) within 90 days prior to consent or during Screening*
* In patients living with HIV: CD4+ T cell count less than 100 cells/mm3 within 90 days prior to consent or during Screening*

  * Indicates an exclusion criterion that may depend on laboratory results and other clinical assessments to be ordered during Screening after confirming the participant is otherwise eligible. If the test was performed as standard-of-care in the 90 days prior to consent, it does not need to be re-done for eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include participants with cirrhosis of the liver.
Sampling Method: Non-Probability Sample
Enrollment: 1222 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2030-10-24 (Estimated); Study Completion 2030-10-24 (Estimated)

PRIMARY OUTCOMES:
Time-to-decompensation | 3 years
  Time-to-decompensation, defined as any of the following events:
  * Ascites: definite as determined by adjudication
  * Hepatic Encephalopathy (HE): definite or highly likely as determined by adjudication
  * Portal hypertensive upper gastrointestinal (GI) bleeding: definite as determined by adjudication

SECONDARY OUTCOMES:
Number of decompensations | 3 years
  Number of decompensations (treated as a count variable in analyses)
All-cause mortality | 3 years
  All-cause mortality (treated as time-to-event in analyses)
Adjudicated liver-related mortality | 3 years
  Adjudicated liver-related mortality (treated as time-to-event in analyses)
All-cause hospitalizations | 3 years
  All-cause hospitalizations (treated as a count variable in analyses)
Number of liver-related hospitalizations | 3 years
  Liver-related hospitalizations (treated as a count variable in analyses)
Time to liver transplantation | 3 years
  Liver transplantation (treated as time-to-event in analyses)
Time to development of hepatocellular carcinoma (HCC) | 3 years
  Development of HCC (treated as time-to-event in analyses)
Time to development of portal and/or mesenteric vein thrombosis | 3 years
  Development of portal and/or mesenteric vein thrombosis (treated as time-to-event in analyses)
Change in liver stiffness as measured by vibration-controlled transient elastography (VCTE) | 3 years
  Liver stiffness as measured by VCTE (treated as continuous measure in analyses)
Degree of fibrosis as measured by fibrosis-4 index (FIB-4) | 3 years
  Degree of fibrosis as measured by FIB-4 (treated as continuous measure in analyses)
Overall physical health and overall mental health as measured by Patient Reported Outcomes Measurement Information System (PROMIS-29+2 profile v2.1) | 3 years
  Overall physical health and overall mental health as measured by Patient Reported Outcomes Measurement Information System (PROMIS-29+2 profile v2.1) relevant "T-scores," a continuous measure. T-scores are normalized to the population and are centered at 50 with anticipated standard deviation of 10. A higher score means better "health."
Change in cognitive function as measured by Stroop Test | 3 years
  Change in cognitive function as measured by Stroop Test (treated as continuous measure in analyses). Measured as time to complete the test. A higher score means longer time to complete, which means more impaired function. Minimum score is 0, and there is no maximum score.
Change in frailty as measured by the Liver Frailty Index | 3 years
  Change in frailty as measured by the Liver Frailty Index (treated as continuous measure in analyses). A higher score means the participant is more frail. The score is based on grip strength, number of chair stands per second, and balance time. https://liverfrailtyindex.ucsf.edu/ Maximum score of 6, and there is no minimum score.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Smith, Principal Investigator — Northwestern University
Locations (14):
- United States (14):
  - University of California San Diego NAFLD Research Center, La Jolla, California
  - Keck Medical Center of USC, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - UCSF/Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - University of Miami Health System, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian/Weill Cornell, New York, New York
  - Columbia University Iriving School of Medicine, New York, New York
  - Duke Liver Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Central Virginia Veterans Healthcare System, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Dataset with National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Repository.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Tapper EB, Goldberg D, Parikh ND, Terrault NA, Welch N, Sharpton S, Hameed B, Khalili M, Stolz A, Verna EC, Brown RS Jr, Sanyal AJ, VanWagner L, Ladner DP, Moylan CA, Diehl AM, Jones PD, Loomba R, Dasarathy S, Simonetto DA, Shah VH, Bajaj JS; LCN Study Group. The Liver Cirrhosis Network Cohort Study: Cirrhosis Definition, Study Population, and Endpoints. Am J Gastroenterol. 2025 Mar 1;120(3):570-575. doi: 10.14309/ajg.0000000000002953. Epub 2024 Jul 17. PMID 39018024
- See also: Information about the study — https://www.lcnstudy.org